CLINICAL TRIAL: NCT02910154
Title: Comprehensive Treatment of Angina in Women With Microvascular Dysfunction - a Proof of Concept Study of the iPower Cohort
Brief Title: Comprehensive Treatment of Angina in Women With Microvascular Dysfunction
Acronym: CORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University Hospital Bispebjerg and Frederiksberg (Other); Cambridge Weight Plan Limited (Industry)
Responsible Party: Principal Investigator, Eva Prescott, Professor, MD, DMSc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CORA; R144 A5460 (Other Grant/Funding Number: Region Hovedstadens Forskningsfond til Sundhedsforskning); H-16032518 (Other: Approval by the National Committee on Health Research Ethics)
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Angina Pectoris; Coronary Microvascular Disease
MeSH Terms: conditions — Angina Pectoris; Microvascular Angina | interventions — Diet; Caloric Restriction; Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weight loss, training, medication (Experimental): The intervention program consists of a comprehensive 24-week treatment period of: 1) Body weight loss without significant loss of muscle mass, through low energy diet combined with 2) Exercise training based on interval training and resistance exercise and 3) Optimal medical treatment for hypertension and hypercholesterolemia (with statin and ACE-inhibition). Further, participants in this allocation group receive nutrition counselling.
  The diet products are sponsored by Cambridge Weight Plan. No persons with interest in Cambridge Weight Plan will take part in the intervention phase, analyzing phase, data processing, or publication of data in this study.
  Interventions: Dietary Supplement: Diet; Behavioral: Training; Drug: Medication (with statin and ACE-inhibition)
- Control (No Intervention): The control group receives 24 weeks of usual care according to guidelines of Danish Cardiology Society. Treatment of angina pectoris in absence of coronary artery disease is normally provided by the patient's general practitioner and does not comprise intensive lifestyle intervention or medical treatment. If control group participants in this study need medical therapy for hypertension or hypercholesterolemia, this will be effectuated by the researcher, MD. Then, control participants will be monitored with blood pressure and LDL blood samples and receive medicine adjustments according to National Prevention Guidelines during the full study period.

INTERVENTIONS:
Dietary Supplement: Diet — Weight loss achieved by following an evidence-based low energy diet of 800-1200 kcal/day for 12 weeks (Cambridge Weight Plan). Hereafter follow 12 weeks of 'weight maintenance' with consumption of normal heart healthy diet. Goal: total weight loss of at least 10% without significant loss of muscle mass. Monitored and supervised by a dietician
  Other Names: Low Energy Diet
  Arms: Weight loss, training, medication
Behavioral: Training — Aerobic interval training and resistance exercise in group sessions twice weekly throughout the 24-week intervention. Training intensity individually adapted to the restricted calorie intake. Goal: Improved VO2 peak (at least 10%). Monitored by a physiotherapist.
  Other Names: Aerobic Exercise Training
  Arms: Weight loss, training, medication
Drug: Medication (with statin and ACE-inhibition) — Medical treatment for hypertension and/or hypercholesterolemia if systolic blood pressure > 130 and/or low density lipoprotein (LDL) > 2.0.
  Other Names: Medical treatment for hypertension and hypercholesterolemia
  Arms: Weight loss, training, medication

SUMMARY:
Angina is the most common symptom of coronary heart disease among women but unlike men most women do not have stenosis of the coronary arteries. In a large proportion of these women, coronary microvascular dysfunction (CMD) is thought to be the cause of angina. However, CMD is also demonstrable in the asymptomatic population, and may merely be an innocent bystander related to the presence of cardiovascular risk factors rather than a cause of angina symptoms.

The aim of this study is to determine whether comprehensive intervention is feasible and results in improvement in both angina and microvascular function in these patients.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction is found to be associated with a significant adverse prognosis. The condition is strongly associated with increased future risk of major cardiovascular events, frequent hospital readmission, continued angina and loss of quality of life compared to the general population.

Pathophysiology of microvessel disease:

In the heart 95% of the blood flow is controlled by the microcirculation. When oxygen demand is increased the normal response of the microvessels is to reduce resistance in order to increase flow. When microvessels are dysfunctional the blood flow in the larger coronary vessels does not increase sufficiently to meet oxygen demand, thus leading to ischemia and pain. The main causes are thought to be dysfunction of endothelium and structural changes such as perivascular fibrosis and changes in vascular smooth muscle cells. In addition to vasodilation the endothelium plays a central role in the atherosclerotic process by generating vasoactive and anticoagulant factors that are important mediators of thrombosis. Coronary microvessel dysfunction (CMD) has been shown to be a strong predictor of poor cardiovascular prognosis in a wide group of cardiac patients.

Rationale for intervention:

In women with angina and no obstructive stenosis of the coronary vessels cardiovascular risk factors are common. Among 3000 Danish women with angina and open arteries, 12% had diabetes, 48% hypertension, 20% were smokers and the mean body mass index was 27 kg/m2. In a randomized trial among overweight patients with coronary artery disease both a large weight loss and intensive exercise training have shown to significantly improve coronary flow velocity reserve (CFVR). Small studies addressing risk factors individually suggest an effect on peripheral vascular function of exercise training, statin therapy, and weight loss. Pre-diabetes is found in eighty percent of these patients and is strongly associated to microvessel disease. Lifestyle intervention significantly reduces risk of developing diabetes. Medical treatment targeting microvessel dysfunction in patients with angina has not been systematically tested but small studies indicate an effect of beta-blockers and Angiotensin Converting Enzyme (ACE)-inhibition on coronary microvessel function. Small studies indicate effect of individual interventions but mainly on the function of peripheral vessels. A comprehensive intervention simultaneously targeting CMD and angina has not previously been attempted.

The rationale for this present intervention is to test this concept in women with angina and CMD.The study is a pilot study which, if successful, will be expanded to a multicentre, intervention trial with prognostic outcome. A large study showing improved prognosis is of crucial importance for treatment of this patient group to become part of guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients will be recruited and included from the ongoing iPower study.(the acronym iPower stands for: improving diagnosis and treatment of women with angina pectoris and microvascular disease)

* Female gender
* 40-75 years of age
* Referred to a cardiac centre for assessment with coronary angiography due to chest pain or other signs of ischemia leaving out ST-segment elevation myocardial Infarction (STEMI) or NSTEMI patients (elevated enzymes, electrocardiographic (ECG) changes/no ECG changes)
* No significant stenotic lesions at the following coronary angiography defined as > 50% stenosis of epicardial vessels. Patients are included within 1 year after coronary angiography.

  * Angina with a symptom burden of symptoms > monthly
  * Impaired coronary microvascular function, defined as a Transthoracic Doppler Echocardiography measured CFVR < 2.5 with a good quality (quality index > 3)
  * BMI > 26 or BMI >= 25 combined with a waist hip ratio of >=0.8
  * Informed consent

Exclusion Criteria:

* Previously verified myocardial infarction, verified in medical records: ST-elevation myocardial infarction, elevated coronary markers or Non ST-elevation myocardial infarction
* Previous percutaneous coronary intervention or coronary artery bypass graft.
* Left ventricular ejection fraction (LVEF) < 45% assessed by echocardiography within 6 months before inclusion
* Any allergies to the content of the low energy diet (gluten/nuts), allergy to dipyridamole, adenosine, or theophyllamine
* Significant valvular heart disease
* Congenital heart disease
* Severe asthma
* Severe chronic obstructive pulmonary disease (COPD): forced expiratory volume in 1st second (FEV1) < 50% of predicted (age, height, ethnicity)
* Severe comorbidity with limited life-expectancy < 1 year
* Chest pain with a strongly suspected non-ischemic etiology (e.g. pericarditis, pneumonia)
* Pregnancy
* Active cancer
* Renal (eGFR < 30) or severe hepatic comorbidity
* Chronic alcohol abuse
* Atrial flutter or fibrillation
* Atrioventricular block > 1st degree
* Diabetes Mellitus type II patients in treatment with Sulphonylureas
* Participation in other trials if relevant for the present study
* Language- or other barrier to giving informed consent
* Physical or mental disabilities contraindicating or hampering diet or exercise training
* Travel distance to research hospital requiring more than 3 hours of travel, making it difficult for the patient to participate

Withdrawal criteria

* Sudden unexpected serious adverse reaction or sustained side effects
* Poor compliance will lead to withdrawal from the study at the mentioned time points: Low energy diet: No weight loss within the first 3 weeks of the intervention period. Medication: < 80% of the prescribed medicine taken within the first 3 weeks. Training: < 50% attendance to training sessions/home training within the first 5 weeks.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-12; Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Changes in coronary microvascular function | Up to 24 months
  Coronary microvascular function will be assessed by transthoracic Doppler stress echocardiography (TTDSE) and measured as Coronary Flow Velocity Reserve (CFVR). CFVR is a measure of microvascular dysfunction in the absence of upstream coronary stenosis. CFVR is the ratio of flow during stress and flow during rest and will be measured with TTDSE of the left anterior descending artery before and during infusion of high dose adenosine (0.14 mg/kg/min).

SECONDARY OUTCOMES:
Changes in symptom burden assessed by the Seattle Angina Questionnaire (SAQ) | Up to 24 months
  The SAQ is a reliable, predictive tool that has been validated in 175 women with a confirmed diagnosis of stable coronary artery disease and angina pectoris. It is a 19-item health-related quality-of-life measure for patients with coronary artery disease. The answers given by the patients in the SAQ's questions are used to calculate scores in five scales: 1. Anginal Stability, 2. Anginal Frequency, 3. Physical Limitation, 4. Treatment Satisfaction and 5) Quality of Life.
  Scale scores are transformed to a 0-100 range by subtracting the lowest possible scale score, dividing by the range of the scale and multiplying by 100. Higher scores indicate less symptom burden. Because each scale monitors a unique dimension of coronary artery disease, no summary score is generated. A score change of 10 points is clinically perceptible to patients and is considered a clinically relevant difference, while a substantial change is considered to be a change of 20 points.
Changes in biomarkers including inflammatory markers and markers of metabolism | Up to 24 months
  Several components in the inflammatory system may be associated with cardiovascular disease and atherosclerosis. A meta-analysis comprising 29 prospective studies associated interleukin-6 (IL6), tumor necrosis factor-alfa (TNF-alfa) and C-reactive protein (CRP) to increased cardiovascular risk independent of traditional risk factors in the healthy population.51
  Fasting blood samples will be collected at baseline and follow-up for assessment of:
  Lipids (total-, low density lipoprotein, very low density lipoprotein, high density lipoprotein, cholesterol and triglycerides), endocrine function (Hba1c, glucose, insulin, thyroid stimulating hormone), kidney function (creatinine, estimated glomerular filtration rate (eGFR)), haematology and inflammatory disease (high sensitive CRP, high sensitive troponin-T, orosomucoid, interleukin-6, tumor necrosis factor alfa (TNF-alfa), adiponectin)
Changes in exercise capacity (VO2peak) | Up to 24 months
  A cardiopulmonary exercise test (CPET) is performed using a bicycle ergometer with breath-by-breath gas exchange measurements (Jaeger, Vyntus CPX, Germany. Participants will be encouraged to continue until exhaustion. Criteria for VO2 peak are levelling off of VO2 despite increasing workload and peak respiratory exchange ratio (peak RER) > 1.10.38 VO2 peak and peak RER are determined at peak effort with 15-second average measurements. VO2 peak is expressed as: VO2 peak (mL/min), VO2 peak (mL/kg body weight/min) and VCO2 peak (mL/min). Predicted VO2 peak is calculated using the equation for sedentary, overweight individuals presented by Wassermann and Hansen. Measured VO2peak in percent of predicted is determined.
Changes in body weight and fat distribution (DEXA scan) | Up to 24 months
  To estimate body composition (body fat mass and fat free mass ) a whole body dual X-ray absorptiometry (DEXA) scan will be performed.
  Body composition will be measured in the morning after a 10-hour fast.
Changes in level of anxiety and depression (HADS questionnaire) | Up to 24 months
  HADS is a self-administered questionnaire consisting of 14 items (each scored 0-3), seven of which concern depression and seven anxiety symptoms. One of the main purposes of this instrument was to identify affective symptoms among somatically ill patients.Therefore, the items focuses on the non-somatic aspects of depression and anxiety, to avoid that symptoms from the somatic disease, such as fatigue, affected the measurements.Depression and anxiety items are summarized separately in two scales ranging from 0 to 21, where a higher score indicates more symptoms.
Changes in systolic and diastolic heart function at rest and during stress including advanced imaging (eg. Strain-Echocardiography) | Up to 24 months
  Diastolic heart function tends to be impaired in obesity and in diabetes, but whether this is also the case in microvessel dysfunction is unclear. Improvement in cardiac function following intervention may be subtle and is more likely measurable during stress. By using global longitudinal and radial 2D strain at rest and during dipyridamole or adenosine stress, we expect that we will be able to detect a smaller difference in myocardial function than by using change in left ventricular ejection fraction (LVEF) assessed by the Simpsons method.
Changes in body weight | Up to 24 months
  Weight in kilograms wil be measured in the morning after a 10-hour fast
changes in hip- and waist circumference | Up to 24 months
  hip and waist circumference will be measured in the morning after a 10-hour fast. Waist circumference is measured halfway between the lower rib and the iliac crest and hip circumference at the maximal gluteal protuberance and calculated as an average of two consecutive measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prescott, MD, DMSc, Principal Investigator — Professor
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Dept. of Cardiology Y builing 67, 1.floor, Bispebjerg Bakke 23, Copenhagen
  - Frederiksberg Hospital, Dept. of Cardiology, Building 16, Y3, Nordre Fasanvej 57, Frederiksberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bairey Merz CN, Shaw LJ, Reis SE, Bittner V, Kelsey SF, Olson M, Johnson BD, Pepine CJ, Mankad S, Sharaf BL, Rogers WJ, Pohost GM, Lerman A, Quyyumi AA, Sopko G; WISE Investigators. Insights from the NHLBI-Sponsored Women's Ischemia Syndrome Evaluation (WISE) Study: Part II: gender differences in presentation, diagnosis, and outcome with regard to gender-based pathophysiology of atherosclerosis and macrovascular and microvascular coronary disease. J Am Coll Cardiol. 2006 Feb 7;47(3 Suppl):S21-9. doi: 10.1016/j.jacc.2004.12.084. PMID 16458167
- [Result] Shaw LJ, Bugiardini R, Merz CN. Women and ischemic heart disease: evolving knowledge. J Am Coll Cardiol. 2009 Oct 20;54(17):1561-75. doi: 10.1016/j.jacc.2009.04.098. PMID 19833255
- [Result] Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, Douglas PS. Low diagnostic yield of elective coronary angiography. N Engl J Med. 2010 Mar 11;362(10):886-95. doi: 10.1056/NEJMoa0907272. PMID 20220183
- [Result] Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, Prescott E. Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J. 2012 Mar;33(6):734-44. doi: 10.1093/eurheartj/ehr331. Epub 2011 Sep 11. PMID 21911339
- [Result] Gulati M, Cooper-DeHoff RM, McClure C, Johnson BD, Shaw LJ, Handberg EM, Zineh I, Kelsey SF, Arnsdorf MF, Black HR, Pepine CJ, Merz CN. Adverse cardiovascular outcomes in women with nonobstructive coronary artery disease: a report from the Women's Ischemia Syndrome Evaluation Study and the St James Women Take Heart Project. Arch Intern Med. 2009 May 11;169(9):843-50. doi: 10.1001/archinternmed.2009.50. PMID 19433695
- [Result] Jespersen L, Abildstrom SZ, Hvelplund A, Galatius S, Madsen JK, Pedersen F, Hojberg S, Prescott E. Symptoms of angina pectoris increase the probability of disability pension and premature exit from the workforce even in the absence of obstructive coronary artery disease. Eur Heart J. 2013 Nov;34(42):3294-303. doi: 10.1093/eurheartj/eht395. Epub 2013 Sep 26. PMID 24071763
- [Result] Jespersen L, Abildstrom SZ, Hvelplund A, Prescott E. Persistent angina: highly prevalent and associated with long-term anxiety, depression, low physical functioning, and quality of life in stable angina pectoris. Clin Res Cardiol. 2013 Aug;102(8):571-81. doi: 10.1007/s00392-013-0568-z. Epub 2013 May 1. PMID 23636227
- [Result] Shaw LJ, Merz CN, Pepine CJ, Reis SE, Bittner V, Kip KE, Kelsey SF, Olson M, Johnson BD, Mankad S, Sharaf BL, Rogers WJ, Pohost GM, Sopko G; Women's Ischemia Syndrome Evaluation (WISE) Investigators. The economic burden of angina in women with suspected ischemic heart disease: results from the National Institutes of Health--National Heart, Lung, and Blood Institute--sponsored Women's Ischemia Syndrome Evaluation. Circulation. 2006 Aug 29;114(9):894-904. doi: 10.1161/CIRCULATIONAHA.105.609990. Epub 2006 Aug 21. PMID 16923752
- [Result] Crea F, Lanza GA. Angina pectoris and normal coronary arteries: cardiac syndrome X. Heart. 2004 Apr;90(4):457-63. doi: 10.1136/hrt.2003.020594. No abstract available. PMID 15020531
- [Result] Bugiardini R, Bairey Merz CN. Angina with "normal" coronary arteries: a changing philosophy. JAMA. 2005 Jan 26;293(4):477-84. doi: 10.1001/jama.293.4.477. PMID 15671433
- [Result] Phan A, Shufelt C, Merz CN. Persistent chest pain and no obstructive coronary artery disease. JAMA. 2009 Apr 8;301(14):1468-74. doi: 10.1001/jama.2009.425. PMID 19351944
- [Result] Cannon RO 3rd. Microvascular angina and the continuing dilemma of chest pain with normal coronary angiograms. J Am Coll Cardiol. 2009 Sep 1;54(10):877-85. doi: 10.1016/j.jacc.2009.03.080. PMID 19712795
- [Result] Sicari R, Rigo F, Cortigiani L, Gherardi S, Galderisi M, Picano E. Additive prognostic value of coronary flow reserve in patients with chest pain syndrome and normal or near-normal coronary arteries. Am J Cardiol. 2009 Mar 1;103(5):626-31. doi: 10.1016/j.amjcard.2008.10.033. Epub 2008 Dec 26. PMID 19231324
- [Result] Pepine CJ, Anderson RD, Sharaf BL, Reis SE, Smith KM, Handberg EM, Johnson BD, Sopko G, Bairey Merz CN. Coronary microvascular reactivity to adenosine predicts adverse outcome in women evaluated for suspected ischemia results from the National Heart, Lung and Blood Institute WISE (Women's Ischemia Syndrome Evaluation) study. J Am Coll Cardiol. 2010 Jun 22;55(25):2825-32. doi: 10.1016/j.jacc.2010.01.054. PMID 20579539
- [Result] Rigo F, Cortigiani L, Pasanisi E, Richieri M, Cutaia V, Celestre M, Raviele A, Picano E. The additional prognostic value of coronary flow reserve on left anterior descending artery in patients with negative stress echo by wall motion criteria. A Transthoracic Vasodilator Stress Echocardiography Study. Am Heart J. 2006 Jan;151(1):124-30. doi: 10.1016/j.ahj.2005.03.008. PMID 16368303
- [Result] Ong P, Athanasiadis A, Borgulya G, Mahrholdt H, Kaski JC, Sechtem U. High prevalence of a pathological response to acetylcholine testing in patients with stable angina pectoris and unobstructed coronary arteries. The ACOVA Study (Abnormal COronary VAsomotion in patients with stable angina and unobstructed coronary arteries). J Am Coll Cardiol. 2012 Feb 14;59(7):655-62. doi: 10.1016/j.jacc.2011.11.015. PMID 22322081
- [Result] Murthy VL, Naya M, Foster CR, Hainer J, Gaber M, Di Carli G, Blankstein R, Dorbala S, Sitek A, Pencina MJ, Di Carli MF. Improved cardiac risk assessment with noninvasive measures of coronary flow reserve. Circulation. 2011 Nov 15;124(20):2215-24. doi: 10.1161/CIRCULATIONAHA.111.050427. Epub 2011 Oct 17. PMID 22007073
- [Result] Pauly DF, Johnson BD, Anderson RD, Handberg EM, Smith KM, Cooper-DeHoff RM, Sopko G, Sharaf BM, Kelsey SF, Merz CN, Pepine CJ. In women with symptoms of cardiac ischemia, nonobstructive coronary arteries, and microvascular dysfunction, angiotensin-converting enzyme inhibition is associated with improved microvascular function: A double-blind randomized study from the National Heart, Lung and Blood Institute Women's Ischemia Syndrome Evaluation (WISE). Am Heart J. 2011 Oct;162(4):678-84. doi: 10.1016/j.ahj.2011.07.011. Epub 2011 Sep 6. PMID 21982660
- [Result] Villano A, Di Franco A, Nerla R, Sestito A, Tarzia P, Lamendola P, Di Monaco A, Sarullo FM, Lanza GA, Crea F. Effects of ivabradine and ranolazine in patients with microvascular angina pectoris. Am J Cardiol. 2013 Jul 1;112(1):8-13. doi: 10.1016/j.amjcard.2013.02.045. Epub 2013 Apr 1. PMID 23558043
- [Result] Pedersen LR, Olsen RH, Frederiksen M, Astrup A, Chabanova E, Hasbak P, Holst JJ, Kjaer A, Newman JW, Walzem R, Wisloff U, Sajadieh A, Haugaard SB, Prescott E. Copenhagen study of overweight patients with coronary artery disease undergoing low energy diet or interval training: the randomized CUT-IT trial protocol. BMC Cardiovasc Disord. 2013 Nov 19;13:106. doi: 10.1186/1471-2261-13-106. PMID 24252596
- [Result] Olsen RH, Pedersen LR, Jurs A, Snoer M, Haugaard SB, Prescott E. A randomised trial comparing the effect of exercise training and weight loss on microvascular function in coronary artery disease. Int J Cardiol. 2015 Apr 15;185:229-35. doi: 10.1016/j.ijcard.2015.03.118. Epub 2015 Mar 11. PMID 25802037
- [Result] Hambrecht R, Wolf A, Gielen S, Linke A, Hofer J, Erbs S, Schoene N, Schuler G. Effect of exercise on coronary endothelial function in patients with coronary artery disease. N Engl J Med. 2000 Feb 17;342(7):454-60. doi: 10.1056/NEJM200002173420702. PMID 10675425
- [Result] Hambrecht R, Walther C, Mobius-Winkler S, Gielen S, Linke A, Conradi K, Erbs S, Kluge R, Kendziorra K, Sabri O, Sick P, Schuler G. Percutaneous coronary angioplasty compared with exercise training in patients with stable coronary artery disease: a randomized trial. Circulation. 2004 Mar 23;109(11):1371-8. doi: 10.1161/01.CIR.0000121360.31954.1F. Epub 2004 Mar 8. PMID 15007010
- [Result] Reriani MK, Dunlay SM, Gupta B, West CP, Rihal CS, Lerman LO, Lerman A. Effects of statins on coronary and peripheral endothelial function in humans: a systematic review and meta-analysis of randomized controlled trials. Eur J Cardiovasc Prev Rehabil. 2011 Oct;18(5):704-16. doi: 10.1177/1741826711398430. Epub 2011 Mar 4. PMID 21450596
- [Result] Kerr SM, Livingstone MB, McCrorie TA, Wallace JM. Endothelial dysfunction associated with obesity and the effect of weight loss interventions. Proc Nutr Soc. 2011 Nov;70(4):418-25. doi: 10.1017/S0029665111001674. Epub 2011 Aug 24. PMID 21861950
- [Result] Diabetes Prevention Program Research Group; Knowler WC, Fowler SE, Hamman RF, Christophi CA, Hoffman HJ, Brenneman AT, Brown-Friday JO, Goldberg R, Venditti E, Nathan DM. 10-year follow-up of diabetes incidence and weight loss in the Diabetes Prevention Program Outcomes Study. Lancet. 2009 Nov 14;374(9702):1677-86. doi: 10.1016/S0140-6736(09)61457-4. Epub 2009 Oct 29. PMID 19878986
- [Result] Galderisi M, D'Errico A. Beta-blockers and coronary flow reserve: the importance of a vasodilatory action. Drugs. 2008;68(5):579-90. doi: 10.2165/00003495-200868050-00002. PMID 18370439
- [Result] Prescott E, Abildstrom SZ, Aziz A, Merz NB, Gustafsson I, Halcox J, Hansen HS, Hansen PR, Kastrup J, Michelsen M, Mygind ND, Ong P, Pena A, Rosengren A, Sechtem U, Sogaard P. Improving diagnosis and treatment of women with angina pectoris and microvascular disease: the iPOWER study design and rationale. Am Heart J. 2014 Apr;167(4):452-8. doi: 10.1016/j.ahj.2014.01.003. Epub 2014 Jan 15. PMID 24655692
- [Result] Leeds AR. Formula food-reducing diets:A new evidence-based addition to the weight management tool box. Nutr Bull. 2014 Sep;39(3):238-246. doi: 10.1111/nbu.12098. PMID 25663817
- [Result] Larsen TM, Dalskov SM, van Baak M, Jebb SA, Papadaki A, Pfeiffer AF, Martinez JA, Handjieva-Darlenska T, Kunesova M, Pihlsgard M, Stender S, Holst C, Saris WH, Astrup A; Diet, Obesity, and Genes (Diogenes) Project. Diets with high or low protein content and glycemic index for weight-loss maintenance. N Engl J Med. 2010 Nov 25;363(22):2102-13. doi: 10.1056/NEJMoa1007137. PMID 21105792
- [Result] Estruch R, Ros E, Salas-Salvado J, Covas MI, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Munoz MA, Sorli JV, Martinez JA, Martinez-Gonzalez MA; PREDIMED Study Investigators. Primary prevention of cardiovascular disease with a Mediterranean diet. N Engl J Med. 2013 Apr 4;368(14):1279-90. doi: 10.1056/NEJMoa1200303. Epub 2013 Feb 25. PMID 23432189 (Retraction: PMID 29897867 N Engl J Med. 2018 Jun 21;378(25):2441-2442)
- [Result] Mygind ND, Michelsen MM, Pena A, Frestad D, Dose N, Aziz A, Faber R, Host N, Gustafsson I, Hansen PR, Hansen HS, Bairey Merz CN, Kastrup J, Prescott E. Coronary Microvascular Function and Cardiovascular Risk Factors in Women With Angina Pectoris and No Obstructive Coronary Artery Disease: The iPOWER Study. J Am Heart Assoc. 2016 Mar 15;5(3):e003064. doi: 10.1161/JAHA.115.003064. PMID 27068634
- [Result] Banerjee S, Peterson LR. Myocardial metabolism and cardiac performance in obesity and insulin resistance. Curr Cardiol Rep. 2007 Apr;9(2):143-9. doi: 10.1007/BF02938341. PMID 17430682
- [Result] Anderson TJ, Uehata A, Gerhard MD, Meredith IT, Knab S, Delagrange D, Lieberman EH, Ganz P, Creager MA, Yeung AC, et al. Close relation of endothelial function in the human coronary and peripheral circulations. J Am Coll Cardiol. 1995 Nov 1;26(5):1235-41. doi: 10.1016/0735-1097(95)00327-4. PMID 7594037
- [Result] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Result] Sasaki S, Higashi Y, Nakagawa K, Kimura M, Noma K, Sasaki S, Hara K, Matsuura H, Goto C, Oshima T, Chayama K. A low-calorie diet improves endothelium-dependent vasodilation in obese patients with essential hypertension. Am J Hypertens. 2002 Apr;15(4 Pt 1):302-9. doi: 10.1016/s0895-7061(01)02322-6. PMID 11991214
- [Result] Guazzi M, Arena R. CardioPulse. New clinical cardiopulmonary exercise testing joint statement from the European Society of Cardiology and American Heart Association. Eur Heart J. 2012 Nov;33(21):2627-8. No abstract available. PMID 23281541
- [Result] Guazzi M, Adams V, Conraads V, Halle M, Mezzani A, Vanhees L, Arena R, Fletcher GF, Forman DE, Kitzman DW, Lavie CJ, Myers J; EACPR; AHA. EACPR/AHA Joint Scientific Statement. Clinical recommendations for cardiopulmonary exercise testing data assessment in specific patient populations. Eur Heart J. 2012 Dec;33(23):2917-27. doi: 10.1093/eurheartj/ehs221. Epub 2012 Sep 5. No abstract available. PMID 22952138
- [Result] VON DOBELN W. Maximal oxygen intake, body size, and total hemoglobin in normal man. Acta Physiol Scand. 1956 Dec 31;38(2):193-9. doi: 10.1111/j.1748-1716.1957.tb01383.x. No abstract available. PMID 13394341
- [Result] Lavie CJ, De Schutter A, Patel DA, Romero-Corral A, Artham SM, Milani RV. Body composition and survival in stable coronary heart disease: impact of lean mass index and body fat in the "obesity paradox". J Am Coll Cardiol. 2012 Oct 9;60(15):1374-80. doi: 10.1016/j.jacc.2012.05.037. Epub 2012 Sep 5. PMID 22958953
- [Result] Beatty AL, Spertus JA, Whooley MA. Frequency of angina pectoris and secondary events in patients with stable coronary heart disease (from the Heart and Soul Study). Am J Cardiol. 2014 Oct 1;114(7):997-1002. doi: 10.1016/j.amjcard.2014.07.009. Epub 2014 Jul 16. PMID 25110069
- [Result] Di Franco A, Villano A, Di Monaco A, Lamendola P, Russo G, Stazi A, Scavone G, Nerla R, Sestito A, Lanza GA, Crea F. Correlation between coronary microvascular function and angina status in patients with stable microvascular angina. Eur Rev Med Pharmacol Sci. 2014;18(3):374-9. PMID 24563437
- [Result] Pedersen LR, Olsen RH, Jurs A, Astrup A, Chabanova E, Simonsen L, Wisloff U, Haugaard SB, Prescott E. A randomised trial comparing weight loss with aerobic exercise in overweight individuals with coronary artery disease: The CUT-IT trial. Eur J Prev Cardiol. 2015 Aug;22(8):1009-17. doi: 10.1177/2047487314545280. Epub 2014 Jul 31. PMID 25082954
- [Result] Kimble LP, Dunbar SB, Weintraub WS, McGuire DB, Fazio S, De AK, Strickland O. The Seattle angina questionnaire: reliability and validity in women with chronic stable angina. Heart Dis. 2002 Jul-Aug;4(4):206-11. doi: 10.1097/00132580-200207000-00002. PMID 12147179
- [Result] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Result] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Result] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Result] Kaptoge S, Seshasai SR, Gao P, Freitag DF, Butterworth AS, Borglykke A, Di Angelantonio E, Gudnason V, Rumley A, Lowe GD, Jorgensen T, Danesh J. Inflammatory cytokines and risk of coronary heart disease: new prospective study and updated meta-analysis. Eur Heart J. 2014 Mar;35(9):578-89. doi: 10.1093/eurheartj/eht367. Epub 2013 Sep 10. PMID 24026779
- [Result] Tsai AG, Wadden TA. The evolution of very-low-calorie diets: an update and meta-analysis. Obesity (Silver Spring). 2006 Aug;14(8):1283-93. doi: 10.1038/oby.2006.146. PMID 16988070